CLINICAL TRIAL: NCT02425033
Title: Endoscopic Submucosal Tunnel Dissection for Endoluminal Partial Myotomy of the Lower Esophageal Sphincter in Patients With Spastic Esophageal Disorders Such as Achalasia
Brief Title: POEM for Spastic Esophageal Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-8327
Record Dates: First submitted 2015-04-02; First posted 2015-04-23 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Esophageal Achalasia
Keywords: POEM; Minimally invasive surgery; Achalasia; Spastic esophageal disorders
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Patients undergoing POEM for spastic esophageal disorders such as achalasia at the University Health Network, Toronto, Canada
  Interventions: Procedure: POEM

INTERVENTIONS:
Procedure: POEM — Under general anesthesia, patient undergoes upper endoscopy and a small longitudinal submucosal incision is created and a dilating balloon is inserted submucosally via the created incision. The balloon is slightly inflated to allow entrance of the endoscope. The gastroscope is advanced into the submucosal space and the tunnel is created via endoscopic or blunt dissection as appropriate. The tunnel is created distally and is stopped several centimeters beyond the lower esophageal sphincter (LES), which can easily be identified using endoscopic landmarks. Using a dissection knife, the clearly visible circular muscles are divided. The longitudinal layer is left intact and the mucosal entry is closed.
  Other Names: Peroral endoscopic myotomy; Endoscopic myotomy

SUMMARY:
This study evaluates the efficacy and safety of the Per-Oral Endoscopic Myotomy (POEM) technique for lower esophageal sphincter myotomy in patients suffering from spastic esophageal disorders such as achalasia at a Canadian institution.

The investigators hypothesize that POEM is a safe and effective technique for the surgical management of such disorders at our institution.

DETAILED DESCRIPTION:
Standard surgical care for spastic esophageal disorders such as achalasia includes a procedure called Heller myotomy.

The treatment in our study, called endoscopic myotomy (also known as peroral endoscopic myotomy - POEM) is different from standard surgery (Heller myotomy) because it is less invasive, is less likely to cause reflux, and usually requires shorter operative times with less loss of blood during the surgery. Although POEM has been adopted worldwide and has proven to be successful, the experience in Canada is very limited to date.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic achalasia or similar spastic esophageal disorder and pre-op barium swallow, manometry, and esophagogastroduodenoscopy being consistent with the diagnosis
* Ability to undergo general anesthesia
* Age > 18 yrs and < 85 yrs. of age
* Ability to give informed consent
* Candidate for elective Heller myotomy

Exclusion Criteria:

* Contraindications for esophagogastroduodenoscopy
* Contraindications for elective Heller myotomy
* BMI > 45
* Currently pregnant
* Refusing to participate in the study or without informed consent
* Concomitant participation in other clinical trial

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of intervention (Symptom severity relief according to pre- and post-operative quality of life questionnaire) | 1 year

SECONDARY OUTCOMES:
Surgical complications | 30 days
  Based on Clavien-Dindo classification of surgical complications
LES pressure (according to manometry) | 6 months
  Lower esophageal sphincter (LES) pressure according to manometry pre and post intervention
pH test (pH level in esophagus) | 6 months
  pre and post intervention
Diameter of the esophageal body | 1 year
  Change in diameter of the esophageal body according to upper endoscopy findings

CONTACTS AND LOCATIONS:
Overall Officials: Eran Shlomovitz, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Result] Pellegrini C, Wetter LA, Patti M, Leichter R, Mussan G, Mori T, Bernstein G, Way L. Thoracoscopic esophagomyotomy. Initial experience with a new approach for the treatment of achalasia. Ann Surg. 1992 Sep;216(3):291-6; discussion 296-9. doi: 10.1097/00000658-199209000-00008. PMID 1417178
- [Result] Ortega JA, Madureri V, Perez L. Endoscopic myotomy in the treatment of achalasia. Gastrointest Endosc. 1980 Feb;26(1):8-10. doi: 10.1016/s0016-5107(80)73249-2. PMID 7358270
- [Result] Inoue H, Minami H, Kobayashi Y, Sato Y, Kaga M, Suzuki M, Satodate H, Odaka N, Itoh H, Kudo S. Peroral endoscopic myotomy (POEM) for esophageal achalasia. Endoscopy. 2010 Apr;42(4):265-71. doi: 10.1055/s-0029-1244080. Epub 2010 Mar 30. PMID 20354937
- [Result] Pasricha PJ, Hawari R, Ahmed I, Chen J, Cotton PB, Hawes RH, Kalloo AN, Kantsevoy SV, Gostout CJ. Submucosal endoscopic esophageal myotomy: a novel experimental approach for the treatment of achalasia. Endoscopy. 2007 Sep;39(9):761-4. doi: 10.1055/s-2007-966764. PMID 17703382
- [Result] Luketich JD, Fernando HC, Christie NA, Buenaventura PO, Keenan RJ, Ikramuddin S, Schauer PR. Outcomes after minimally invasive esophagomyotomy. Ann Thorac Surg. 2001 Dec;72(6):1909-12; discussion 1912-3. doi: 10.1016/s0003-4975(01)03127-7. PMID 11789770
- [Result] Hungness ES, Teitelbaum EN, Santos BF, Arafat FO, Pandolfino JE, Kahrilas PJ, Soper NJ. Comparison of perioperative outcomes between peroral esophageal myotomy (POEM) and laparoscopic Heller myotomy. J Gastrointest Surg. 2013 Feb;17(2):228-35. doi: 10.1007/s11605-012-2030-3. Epub 2012 Sep 28. PMID 23054897
- [Result] Minami H, Isomoto H, Yamaguchi N, Matsushima K, Akazawa Y, Ohnita K, Takeshima F, Inoue H, Nakao K. Peroral endoscopic myotomy for esophageal achalasia: clinical impact of 28 cases. Dig Endosc. 2014 Jan;26(1):43-51. doi: 10.1111/den.12086. Epub 2013 Apr 14. PMID 23581563
- [Result] Pescarus R, Shlomovitz E, Swanstrom LL. Per-oral endoscopic myotomy (POEM) for esophageal achalasia. Curr Gastroenterol Rep. 2014 Jan;16(1):369. doi: 10.1007/s11894-013-0369-6. PMID 24362953
- [Result] Kumta NA, Mehta S, Kedia P, Weaver K, Sharaiha RZ, Fukami N, Minami H, Casas F, Gaidhane M, Lambroza A, Kahaleh M. Peroral endoscopic myotomy: establishing a new program. Clin Endosc. 2014 Sep;47(5):389-97. doi: 10.5946/ce.2014.47.5.389. Epub 2014 Sep 30. PMID 25324996
- [Result] Sharata AM, Dunst CM, Pescarus R, Shlomovitz E, Wille AJ, Reavis KM, Swanstrom LL. Peroral endoscopic myotomy (POEM) for esophageal primary motility disorders: analysis of 100 consecutive patients. J Gastrointest Surg. 2015 Jan;19(1):161-70; discussion 170. doi: 10.1007/s11605-014-2610-5. Epub 2014 Sep 3. PMID 25183406
- [Result] Von Renteln D, Fuchs KH, Fockens P, Bauerfeind P, Vassiliou MC, Werner YB, Fried G, Breithaupt W, Heinrich H, Bredenoord AJ, Kersten JF, Verlaan T, Trevisonno M, Rosch T. Peroral endoscopic myotomy for the treatment of achalasia: an international prospective multicenter study. Gastroenterology. 2013 Aug;145(2):309-11.e1-3. doi: 10.1053/j.gastro.2013.04.057. Epub 2013 May 9. PMID 23665071
- [Result] Saleem AM, Hennessey H, von Renteln D, Vassiliou MC. Atrial fibrillation as an unexpected complication after peroral endoscopic myotomy (POEM): a case report. Surg Laparosc Endosc Percutan Tech. 2014 Oct;24(5):e196-9. doi: 10.1097/SLE.0000000000000094. PMID 25222714
- [Result] Yang D, Wagh MS. Peroral endoscopic myotomy for the treatment of achalasia: an analysis. Diagn Ther Endosc. 2013;2013:389596. doi: 10.1155/2013/389596. Epub 2013 Oct 27. PMID 24282373
- [Result] Ren Z, Zhong Y, Zhou P, Xu M, Cai M, Li L, Shi Q, Yao L. Perioperative management and treatment for complications during and after peroral endoscopic myotomy (POEM) for esophageal achalasia (EA) (data from 119 cases). Surg Endosc. 2012 Nov;26(11):3267-72. doi: 10.1007/s00464-012-2336-y. Epub 2012 May 19. PMID 22609984
- [Result] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542